CLINICAL TRIAL: NCT00264381
Title: Management of Superficial Thrombophlebitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10341; ORA-20030415 (Other: University of Oklahoma Office of Research Administration)
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Superficial Thrombophlebitis; Upper Extremity Superficial Thrombophlebitis; Lower Extremity Superficial Thrombophlebitis
Keywords: Superficial Thrombophlebitis; STP; Fragmin; Ibuprofen; Superficial Thrombus; Superficial Phlebitis; phlebitis
MeSH Terms: conditions — Phlebitis | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibuprofen (Active Comparator): Ibuprofen 800mg tid X 7 days + additional 7 days determined by protocol
  Interventions: Drug: Dalteparin sodium injection

INTERVENTIONS:
Drug: Dalteparin sodium injection — Experimental group: dalteparin sodium 200units/kg subcutaneous on day one, followed by 10,000 units subcutaneous daily for six days plus placebo tablets taken orally three times daily for seven days. Control group: Ibuprofen 800mg orally three times daily for seven days plus placebo injection subcutaneous daily for seven days.
  Other Names: Fragmin

SUMMARY:
The purpose of this study is to test the hypothesis that Fragmin (dalteparin sodium) subcutaneously once daily for 7 days is more effective than Ibuprofen given orally three times daily for 7 days for the treatment of superficial thrombophlebitis (STP).

DETAILED DESCRIPTION:
Superficial thrombophlebitis is a common problem and is thought to affect up to 20% of patients with varicose veins. In the absence of treatment, STP may cause its greatest morbidity with extension of thrombus into the deep venous system and resultant risk of pulmonary embolism.

Current standard therapy for STP consists of local heat, elevation of the extremity, and non-steroidal anti-inflammatory medication. However, no study to date has adequately evaluated the effectiveness of this therapy despite persistence and recurrence of symptoms of STP in many patients.

The purpose of this study is to document the outcome of patients with objectively documented STP who are treated with NSAID therapy (standard care) verses those treated with low-molecular weight heparin (dalteparin sodium) according to a pre-defined treatment regimen.

All patients with documented upper or lower STP will be screened. Each will have a complete baseline and risk factor assessment.

All patients will be randomized in one of two treatment groups:

(a) Experimental group who will receive Fragmin (dalteparin)fixed dose subcutaneously daily for 7 days or (b) Control group who will receive ibuprofen 800mg given orally three times daily for 7 days. All patients will receive study drug for a period of 1-2 weeks with reassessment of STP by ultrasound.

All patients will participate for a period of 3 months with follow up visits at 7-9, and 14-16 day, and 1,3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed upper or lower extremity superficial thrombophlebitis by ultrasound imaging

Exclusion Criteria:

* Active, clinically significant bleeding
* Known hypersensitivity to NSAIDS, heparin or derivatives
* Currently pregnant or < 1 week post-partum
* Acquired bleeding diathesis
* Known inherited bleeding disorder
* Renal failure
* Extremes of weight
* unable to return for repeat diagnostic testing or follow-up visit
* Concurrent deep-vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-10; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Rathbun, M.D., Principal Investigator — University of Oklahoma Medicine/Cardiovascular Section
Locations (2):
- United States (2):
  - Department of Veterans Affairs Medical Center, Oklahoma City, Oklahoma
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Rathbun SW, Aston CE, Whitsett TL. A randomized trial of dalteparin compared with ibuprofen for the treatment of superficial thrombophlebitis. J Thromb Haemost. 2012 May;10(5):833-9. doi: 10.1111/j.1538-7836.2012.04669.x. PMID 22360152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients, inpatient and outpatient, with ultrasound confirmed superficial thrombophlebitis of the upper or lower extremity
Pre-assignment Details: Exclusion criteria: receiving anticoagulant therapy for more than 24 hours, concurrent DVT, active bleeding, hypersensitivity to NSAIDS, pregnant or <1 week post-partum, history of bleeding gastric ulcers, hemorrhagic CVA in last year, platelet count<100K, bleeding disorder, serum creatine > 2mg/dl, BP > 180/110, weight <40kg or >135kg
Groups:
- Ibuprofen 800 mg Tid: Ibuprofen 800mg orally tid for 7 days + one placebo injection daily for 7 days
  + additional 7 days of same therapy based on result of ultrasound at day 7
- Dalteparin 200 U/kg Then 10,000 U Daily: Dalteparin 200 units/kg subcutaneously injection on day one then 10,000 units daily for 6 additional doses + placebo orally for 7 days
  + additional 7 days of same therapy based on results of ultrasound at day 7
Period: Overall Study
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily
Started | 35 | 37
Completed | 35 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily | Total
Number analyzed (Participants) | 35 | 37 | 72
Age Continuous [Mean (Full Range); unit: years] | 52 [19 to 85] | 51 [28 to 88] | 51 [19 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72

OUTCOME MEASURES:

1. Secondary Outcome: Major and Minor Bleeding Secondary to Dalteparin and Ibuprofen Treatment During the 3 Month Follow up.
Description: Number of participants with bleeding events related to treatment
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily
Number analyzed (Participants) | 35 | 37
participants | 0 | 0

2. Primary Outcome: Thrombosis Progression and Venous Thromboembolism (VTE)
Description: Thrombosis progression and deep vein thrombosis at day 14 by ultrasound testing
Time Frame: Day 14
Population: Total number available for follow up
Measure: Number; unit: participants
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily
Number analyzed (Participants) | 35 | 37
participants
  Thrombosis progression | 4 | 0
  VTE | 0 | 0

3. Primary Outcome: Thrombosis Progression or Venous Thromboembolism (VTE) at 3 Months
Description: Symptomatic thrombosis extension (DVT) or pulmonary embolism at 3 months documented by radiologic testing.
Time Frame: 3 months
Population: Participants available for follow up
Measure: Number; unit: participants
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily
Number analyzed (Participants) | 35 | 37
participants
  Thrombosis progression | 6 | 4
  VTE | 0 | 1

4. Secondary Outcome: Change From Baseline to Day 14 in Pain Assessment
Description: Change in pain at day 14 as measured by 11-point Box Pain Scale, 0 being the least amount of pain, and 10 the most amount of pain
Time Frame: Day 1, Day 14
Population: Participants available at follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily
Number analyzed (Participants) | 35 | 37
units on a scale | -2.28 (2.69) | -2.23 (2.01)

ADVERSE EVENTS:
Arm/Group | Ibuprofen 800 mg Tid | Dalteparin 200 U/kg Then 10,000 U Daily
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/37
Other Adverse Events (participants affected / at risk) | 1/35 | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen 800 mg Tid (N=35) | Dalteparin 200 U/kg Then 10,000 U Daily (N=37)
Major bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Not related to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen 800 mg Tid (N=35) | Dalteparin 200 U/kg Then 10,000 U Daily (N=37)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No